CLINICAL TRIAL: NCT00654537
Title: A 6 Week Open Label, Dose Comparison Study to Evaluate the Safety and Efficacy of Rosuvastatin Versus Atorvastatin, Pravastatin, and Simvastatin in Subjects With Hypercholesterolemia.
Brief Title: STELLAR-Rosuvastatin vs. Atorvastatin, Pravastatin, Simvastatin Across Dose Ranges
Acronym: STELLAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Elisabeth Björk, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4522IL/0065; D3560C00065
Record Dates: First submitted 2008-04-03; First posted 2008-04-08 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Hypercholesterolemia
Keywords: Cholesterol; hypercholesterolemia; low density lipoproteins
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium; Atorvastatin; Pravastatin; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Rosuvastatin
  Interventions: Drug: Rosuvastatin
- 2 (Active Comparator): Atorvastatin
  Interventions: Drug: Atorvastatin
- 3 (Active Comparator): Pravastatin
  Interventions: Drug: Pravastatin
- 4 (Active Comparator): Simvastatin
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Rosuvastatin
  Other Names: Crestor
  Arms: 1
Drug: Atorvastatin
  Other Names: Lipitor
  Arms: 2
Drug: Pravastatin
  Other Names: Lipostat
  Arms: 3
Drug: Simvastatin
  Other Names: Zocor
  Arms: 4

SUMMARY:
To compare the efficacy of various doses of rosuvastatin with atorvastatin, pravastatin & simvastatin in reducing levels of low density lipoprotein cholesterol in subjects with hypercholesterolaemia.

ELIGIBILITY:
Inclusion Criteria:

* Discontinuation of all previous lipid lowering therapy.
* Fasting LDL-c levels of between 160mg/dl - 250 mg/dl at Visits 2 & 3 for subjects not on lipid lowering therapy at Visit 1.
* Other lipid parameters as specified in the protocol.

Exclusion Criteria:

* The use of lipid lowering drugs or dietary supplements after Visit 1.
* Active arterial disease eg Unstable angina, or recent arterial surgery
* Abnormal laboratory parameters as defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5625 (Estimated)
Dates: Start 2001-04; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Percentage change in low density lipoprotein cholesterol. | 4 & 6 weeks

SECONDARY OUTCOMES:
Percentage change in other lipid parameters as defined by the protocol | 6 weeks
Safety evaluation | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Miller, MD, Study Director — AstraZeneca; Russell Esterline, Study Chair — AstraZeneca